CLINICAL TRIAL: NCT00856739
Title: Obesity and Initiation of Osteoarthritis
Brief Title: Obesity and the Initiation of Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: A6650-R; 7924 (Other: IRB protocol number)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: obesity; arthritis
MeSH Terms: conditions — Obesity; Arthritis

STUDY DESIGN:
Observational Model: Ecologic or Community
Biospecimen Retention: Samples Without DNA — One tube of blood identified with a unique number.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Healthy adults aged 20-60 of varying weights will participate in this minimally invasive study. There is one 4-hour appointment for which subjects are paid $120. The tests involve: 1 tube blood draw, 1 gait test (motion capture) and 1 MR of both knees.

DETAILED DESCRIPTION:
The tests will be done at the VA and Stanford and are not dangerous or painful. They are designed to help us learn more about the relationship of excess weight on cartilage degradation by testing a biomarker in blood. Gait testing involves walking in a lab that is about 20 meters long about 20 times. MR involves lying in a tube for less than 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults aged 20-60 who have no history of LE surgery
* Healthy adults able to walk 30 minutes
* Healthy adults able to have MR

Exclusion Criteria:

* Adults who have had LE surgery
* Adults cannot walk 30 minutes
* Adults who cannot tolerate MR
* Adults with osteoarthritis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults aged 20-60, of varying weights.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P. Andriacchi, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Result] Blazek K, Favre J, Asay J, Erhart-Hledik J, Andriacchi T. Age and obesity alter the relationship between femoral articular cartilage thickness and ambulatory loads in individuals without osteoarthritis. J Orthop Res. 2014 Mar;32(3):394-402. doi: 10.1002/jor.22530. Epub 2013 Nov 26. PMID 24281940
- [Result] Blazek K, Asay JL, Erhart-Hledik J, Andriacchi T. Adduction moment increases with age in healthy obese individuals. J Orthop Res. 2013 Sep;31(9):1414-22. doi: 10.1002/jor.22390. Epub 2013 Jun 4. PMID 23737249

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Weight: Body mass index between 18 and 25 kg/m^2
- Overweight: Body mass index between 25 and 30 kg/m^2
- Obese: Body mass index over 30 kg/m^2
Period: Overall Study
Arm/Group | Normal Weight | Overweight | Obese
Started | 70 | 52 | 55
Completed | 70 | 52 | 55
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: no self-reported chronic pain or significant injury in any of the lower extremity joints or lower back
Groups:
- Normal Weight: Body mass index between 18 and 25 kg/m^2, no self-reported chronic pain or significant injury in any of the lower extremity joints or lower back
- Overweight: Body mass index between 25 and 30 kg/m^2, no self-reported chronic pain or significant injury in any of the lower extremity joints or lower back
- Obese: Body mass index between 30 and 50 kg/m^2, no self-reported chronic pain or significant injury in any of the lower extremity joints or lower back
- Total: Total of all reporting groups
Arm/Group | Normal Weight | Overweight | Obese | Total
Number analyzed (Participants) | 70 | 52 | 55 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (11.99) | 40.91 (13.08) | 39.8 (11.27) | 39.89 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 16 | 34 | 90
  Male | 30 | 36 | 21 | 87

OUTCOME MEASURES:

1. Primary Outcome: Gait Knee Adduction Moment
Time Frame: baseline or first and only visit.
Population: Obese were compared to healthy weight subjects. No overweight subjects were used in this analysis. Subjects were excluded based on MRI evidence of cartilage defects, osteophytes, ligament tears, meniscal tears, or bone marrow edema.
Measure: Mean (Standard Deviation); unit: percent body weight (N)*height (m)
Arm/Group | Normal Weight | Obese
Number analyzed (Participants) | 59 | 36
percent body weight (N)*height (m) | 3.14 (0.816) | 2.39 (0.765)

2. Primary Outcome: Cartilage Thickness
Description: Medial/lateral thickness ratio
Time Frame: baseline or first and only visit.
Population: Overweight and obese were combined based on similarities found in literature. Subjects were excluded based on MRI evidence of cartilage defects, osteophytes, ligament tears, meniscal tears, or bone marrow edema.
Measure: Mean (Standard Deviation); unit: mm/mm
Groups:
- Normal Weight Young: Body mass index between 18 and 25 kg/m^2, age between 20 and 35
- Overweight and Obese Young: Body mass index between 27 and 50 kg/m^2, age between 20 and 35
- Normal Weight Middle Age: Body mass index between 18 and 25 kg/m^2, age between 35 and 60
- Overweight and Obese Middle Age: Body mass index between 27 and 50 kg/m^2, age between 35 and 60
Arm/Group | Normal Weight Young | Overweight and Obese Young | Normal Weight Middle Age | Overweight and Obese Middle Age
Number analyzed (Participants) | 28 | 28 | 27 | 27
mm/mm | 1.069 (0.097) | 1.04571 (0.169) | 1.051 (0.127) | 1.069 (0.139)

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed.
Groups:
- Obese: Body mass index between 30 and 50 kg/m^2
Arm/Group | Normal Weight | Overweight | Obese
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes